CLINICAL TRIAL: NCT02700334
Title: Effect of Dapagliflozin on Insulin Secretion and Insulin Sensitivity in Patients With Prediabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, Researcher Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAPA-PREDIABETES
Record Dates: First submitted 2016-02-23; First posted 2016-03-07 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Prediabetes; Impaired Fasting Glucose; Impaired Glucose Tolerance
Keywords: Prediabetes; Impaired fasting glucose; Hyperglycemia; Impaired glucose tolerance; Glucose intolerance; Dapagliflozin; Sodium glucose cotransporter 2 inhibitor; SGLT2
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Hyperglycemia | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin capsules, 10 mg, one per day before breakfast during 12 weeks.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo capsules, one per day before breakfast during 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg, one per day before breakfast during 12 weeks.
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Placebo — one per day before breakfast during 12 weeks.
  Other Names: Calcined magnesium
  Arms: Placebo

SUMMARY:
Prediabetes is a term that refers to alterations in glucose homeostasis, including impaired fasting glucose (IFG), impaired glucose tolerance (IGT) or both, involving a higher risk of progression type 2 diabetes mellitus (T2DM).

Dapagliflozin is a selective and reversible inhibitor of sodium-glucose type 2 (SGLT-2) co-transporter, which reduces renal glucose reabsorption and promotes the glucose excretion through urine, so that the blood glucose is improved in patients with T2DM. Although this mechanism is independent of insulin, there are evidence of improved secretion and insulin sensitivity, so it is interesting to assess these effects in patients with prediabetes, as potential therapy for treating such disorders and prevent progression to T2DM.

The aim of this study is to evaluate the effect of Dapagliflozin on insulin secretion and insulin sensitivity in patients with prediabetes.

The investigators hypothesis is that the administration of dapagliflozin improve insulin secretion and insulin sensitivity in patients with prediabetes.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial in 24 patients with a diagnosis of prediabetes in accordance with the American Diabetes Association (ADA) without treatment.

They will be assigned randomly two groups of 12 patients each to receive 10 mg of Dapagliflozin (Forxiga, Astra Zeneca) or placebo, one per day before breakfast during 12 weeks.

There will be calculated Area Under the Curve of glucose and insulin, total insulin secretion (Insulinogenic index), first-phase of insulin secretion (Stumvoll index) and insulin sensitivity (Matsuda index).

This protocol it's already approved by the local ethics committee and written informed consent it's going to be obtained from all volunteers.

Statistical analysis will be presented through measures of central tendency and dispersion, average and deviation standard for quantitative variables; frequencies and percentages for variable qualitative. Qualitative variables will be analyzed by X2, will be used for differences inter-group Mann-Whitney U Test and Wilcoxon Test for the within-groups differences. It will be considered statistical significance p ≤0.05.

This protocol was approved by a local ethics committee and written informed consent will be obtained from all volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Patients both sexes
* Age between 30 and 60 years
* Diagnosis of prediabetes according ADA criteria (fasting blood glucose levels between 100-126 mg/dl; postprandial blood glucose levels after an oral glucose tolerance test with 75 of oral glucose between 140-199 mg/dl; or glycosylated hemoglobin between 5.7-6.4%)
* Informed consent signed

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Hypersensibility to ingredients of intervention
* Physical impossibility for taking pills
* Known uncontrolled renal, hepatic, heart or thyroid diseased
* Diabetes diagnosis
* Previous treatment for glucose
* Body Mass Index ≥35 kg/m2
* Triglycerides ≥500 mg/dL
* Total cholesterol ≥240 mg/dL
* Low density lipoprotein (c-LDL) ≥190 mg/dL
* Blood Pressure ≥140/90 mmHg

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MANUEL GONZALEZ, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Intstituto de Terapeútica Experimental y Clínica. Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dapagliflozin | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (6.3) | 46.7 (9.8) | 49.1 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 24
Fasting Glucose [Mean (Standard Deviation); unit: mmol/L] | 5.9 (0.4) | 6.0 (0.4) | 6.0 (0.4)
Postprandial Glucose [Mean (Standard Deviation); unit: mmol/L] | 9.2 (1.4) | 9.5 (1.4) | 9.4 (1.4)
First Phase of Insulin Secretion [Mean (Standard Deviation); unit: index] — Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the first phase of insulin secretion
  index | 1126 (604) | 1708 (709) | 1417 (656.5)
Total Insulin Secretion [Mean (Standard Deviation); unit: index] — The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔABC insulin/ΔABC glucose), the entered values reflect the total insulin secretion
  index | 0.69 (0.31) | 0.49 (0.17) | 0.6 (0.2)
Insulin Sensitivity [Mean (Standard Deviation); unit: index] — Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
  index | 1.78 (1.09) | 1.94 (0.72) | 1.9 (0.9)
Glycosylated Hemoglobin [Mean (Standard Deviation); unit: percentage] | 5.8 (0.3) | 5.8 (0.5) | 5.8 (0.4)
Body Weight [Mean (Standard Deviation); unit: kg] | 80.8 (16.3) | 83.5 (8.2) | 82.2 (12.3)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.3 (3.5) | 33.0 (2.2) | 31.7 (2.9)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 5.0 (0.9) | 4.7 (0.6) | 4.9 (0.8)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 1.5 (0.5) | 1.4 (0.6) | 1.5 (0.6)
High Density Lipoprotein cholesterol (HDL-c) [Mean (Standard Deviation); unit: mmol/L] | 1.6 (0.2) | 1.5 (0.2) | 1.6 (0.2)
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: IU/L] | 33.3 (16.0) | 37.1 (26.8) | 35.2 (21.4)
Aspartate Aminotransferase (AST) [Mean (Standard Deviation); unit: IU/L] | 36.0 (8.0) | 32.7 (19.6) | 34.4 (13.8)
Creatinine [Mean (Standard Deviation); unit: mmol/L] | 0.06 (0.01) | 0.07 (0.02) | 0.07 (0.02)
Uric Acid [Mean (Standard Deviation); unit: μmol/L] | 334 (70) | 312 (101) | 323 (85.5)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 124 (9) | 126 (11) | 125 (10)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 78 (10) | 77 (11) | 78 (11)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Glucose
Description: The fasting glucose levels will be evaluated with enzymatic/colorimetric techniques and the entered values reflect the fasting glucose level at week 12
Time Frame: Fasting Glucose levels at week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 5.1 (0.3) | 5.9 (0.5)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.005, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Postprandial Glucose
Description: Postprandial glucose will be evaluated after a oral glucose tolerance test with enzymatic/colorimetric techniques and the entered values reflect the insulin sensitivity at week 12
Time Frame: Postprandial Glucose levels at Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 8.4 (1.5) | 8.7 (2.7)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.093, Wilcoxon (Mann-Whitney)

3. Primary Outcome: First Phase of Insulin Secretion
Description: The first phase of insulin secretion will be calculated with Stumvoll index and the entered values reflect the frst phase of insulin secretion at week 12. Human studies support the critical physiologic role of the first-phase of insulin secretion in the maintenance of postmeal glucose homeostasis.
  First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), the entered values reflect the first phase of insulin secretion
Time Frame: First Phase of Insulin Secretion at Week 12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
index | 1096 (388) | 1379 (566)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.878, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Total Insulin Secretion
Description: Total insulin secretion will be calculated with insulinogenic index and the entered values reflect the total insulin secretion at week 12.
  The insulinogenic index is a ratio that relates enhancement of circulating insulin to the magnitude of the corresponding glycemic stimulus.
  Total insulin secretion was calculated with the insulinogenic index (ΔABC insulin/ΔABC glucose), the entered values reflect the total insulin secretion
Time Frame: Total Insulin Secretion at Week 12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
index | 0.50 (0.18) | 0.67 (0.33)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.959, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Insulin Sensitivity
Description: Insulin sensitivity will be calculated with Matsuda index and the entered values reflect the insulin sensitivity at week 12.
  Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
Time Frame: Insulin Sensitivity at Week 12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
index | 2.63 (1.04) | 1.94 (0.71)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.005, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Glycosylated Hemoglobin
Description: Glycosylated hemoglobin will be evaluated by ELISA and the entered values reflect the glycosylated hemoglobin at week 12
Time Frame: Glycosylated Hemoglobin at Week 12
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
percentage | 5.7 (0.3) | 5.9 (0.4)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.331, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Body Weight
Description: The body weight will be measured with a bioimpedance balance and the entered values reflect the body weight at week 12
Time Frame: Body Weight at Week 12
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
kg | 77.8 (14.9) | 82.5 (7.5)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.005, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Body Mass Index
Description: Body Mas Index will be calculated with the Quetelet index formula and the entered values reflect the body mass index at week 12
Time Frame: Body Mass Index at Week 12
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
kg/m^2 | 29.2 (3.1) | 32.6 (2.3)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.005, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Total Cholesterol
Description: Total cholesterol levels will be evaluated by enzymatic/colorimetric techniques and the entered values reflect the total cholesterol level at week 12
Time Frame: Total Cholesterol levels at Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 4.8 (0.9) | 4.7 (0.8)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.575, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Triglycerides
Description: Triglycerides levels will be evaluated with enzymatic/colorimetric techniques and the entered values reflect the triglycerides level at week 12
Time Frame: Triglycerides levels at Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 1.5 (0.7) | 1.6 (0.2)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.314, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: High Density Lipoprotein Cholesterol (HDL-c)
Description: HDL-c levels will be evaluated with enzymatic/colorimetric techniques and the entered values reflect the c-HDL level at week 12
Time Frame: HDL-c levels at Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 1.5 (0.7) | 1.6 (0.2)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.721, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: ALT levels will be evaluated with enzymatic/colorimetric techniques at week 12
Time Frame: ALT levels at Week 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
IU/L | 29.3 (13.6) | 27.7 (14.0)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.066, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Aspartate Aminotransferase (AST)
Description: AST levels will be evaluated with enzymatic/colorimetric techniques at week 12
Time Frame: AST levels at Week 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
IU/L | 29.3 (13.6) | 27.7 (14.0)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.333, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Creatinine
Description: Creatinine levels will be evaluated with enzymatic/colorimetric techniques at week 12
Time Frame: Creatinine levels at Week 12
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
µmol/L | 79.6 (35.4) | 61.9 (17.7)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.859, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Uric Acid
Description: Uric acid levels will be evaluated with enzymatic/colorimetric techniques at week 12
Time Frame: Uric Acid levels at Week 12
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
µmol/L | 261.7 (59.5) | 303.4 (83.3)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.009, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Systolic Blood Pressure
Description: Systolic Blood pressure will be measured with a digital sphygmomanometer and the entered values reflect the blood pressure at week 12
Time Frame: Systolic Blood Pressure at Week 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
mmHg | 124 (12) | 123 (12)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.919, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Diastolic Blood Pressure
Description: as for outcome 16
Time Frame: Diastolic Blood Pressure at Week 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 12 | 12
mmHg | 77 (10) | 74 (10)
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; Test type: Other; p = 0.720, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study (12 weeks)
Arm/Group | Dapagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 7/12 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin (N=12) | Placebo (N=12)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Edema in upper extremities (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes